CLINICAL TRIAL: NCT05068076
Title: Role of Kupffer Phase Specific Ultrasound Contrast Agent (Perfluorobutane) in Lesion Detection, Targeting and Response Assessment for Ablation Therapy (Radiofrequency/ Microwave Ablation) of Hepatocellular Carcinoma
Brief Title: Role of Perfluorobutane in Lesion Detection, Targeting and Response Assessment for Ablation of HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ILBS-HCC-04
Record Dates: First submitted 2021-09-08; First posted 2021-10-05 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma; Microwave Ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — perfluorobutane; Sonazoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing ablation for HCC (Experimental): Pre-procedure CEUS will be performed on patients undergoing ablation followed by targeting of lesions for precise needle placement in the Kupffer phase. 2 hours post procedure USG with contrast will also be done for response assessment
  Interventions: Drug: Perfluorobutane

INTERVENTIONS:
Drug: Perfluorobutane — Perfluorobutane enhanced ultrasound will be done prior to ablation of HCC and after 2hours post ablation and comparison will be done with 1 month post procedure CT/MRI
  Other Names: Sonazoid

SUMMARY:
Primary liver cancers are the sixth most common malignancies worldwide, with hepatocellular carcinoma (HCC) accounting for approximately 80% of them. The Barcelona Clinic Liver Cancer (BCLC) classification is widely used in the management of HCC. At the time of diagnosis, fewer than 30% of the patients qualify for resection or transplant due to the large size or multiplicity of the lesions, background chronic liver disease, and other comorbidities.

However, the recent spread of surveillance has led to early detection of hepatocellular carcinoma (HCC), and the chance of receiving local treatment has increased. There are several options to treat small HCCs, including surgical resection, chemical ablation, transplantation, and percutaneous ablation (RFA/MWA).

Today, percutaneous ablation plays a key role in the treatment of early-stage HCC because it is less invasive than surgical resection and has a good efficacy. However, targeting of lesions under USG alone may be misleading as there may be an enhancing component which is not seen on plain ultrasound. To overcome this problem contrast enhanced ultrasound may be used intra-procedurally, however conventional ultrasound contrast agents show washout by 5 minutes from the system.

In this study, the investigators prospectively analyze patients undergoing ablation with the help of precise needle placement using a Kupffer phase ultrasound contrast agent (perfluorobutane) and their post procedure response assessment.

DETAILED DESCRIPTION:
International status:

Hepatocellular carcinoma (HCC) is the most common primary malignancy of the liver with increasing incidence due to hepatitis B and C viruses . Ultrasound (USG) with, or without alpha feto-protein levels is a standard tool for surveillance of HCC. However, it leads to suboptimal detection rate and false referrals in the US . Use of an ultrasound contrast agent can be helpful in surveillance and diagnosis of focal liver lesions . Second generation ultrasound contrast agents like sulfur hexafluoride (SonoVue), perflutren lipid (Definity) and perfluorobutane (Sonazoid) are microbubbles composed of a phospholipid shell encompassing a low-solubility gas . The characteristic property of Sonazoid is its ability to accumulate in the reticuloendothelial system (such as the Kupffer cells in the liver) for a sustained period of time (up to 60 mins), which is not seen with other second generation contrast agents . Malignant liver lesions do not contain Kupffer cells so these lesions appear hypoechoic in the Kupffer phase (10-60 minutes) .

CEUS has been previously used for targeting of lesions for radiofrequency ablation, however the contrast agent used in the study was Definity . CEUS with Sonazoid has been frequently used in Japan, South Korea and Norway for diagnosis and surveillance. Diagnosis with Sonazoid involves the vascular phase (10 sec to 5 minutes) and the Kupffer phase (10-60 minutes). The vascular phase shows the tumor vascularity and the Kupffer phase shows the absence of reticuloendothelial cells in the lesion (2-4). In case of a new lesion detected in the Kupffer phase or a doubt regarding a previously detected lesion, defect reperfusion imaging can be done for confirmation and diagnosis . In a comparison between SonoVue and Sonazoid in diagnosis of liver lesions, Sonazoid was not inferior to SonoVue in diagnosis and significantly better in detecting lesions during whole liver scanning .

A study was done using Sonazoid enhanced ultrasound for targeting lesions not detected by conventional USG for ablation therapy, and it was found that CEUS detected 97% of the viable tumours compared to 83% by conventional USG. Furthermore, 93% of the lesions which were not detected on conventional USG were treated successfully using late phase of the contrast agent as a guiding tool . However, CEUS using Sonazoid was not used to assess treatment response in this study. A meta-analysis assessing the treatment response after radiofrequency ablation of HCC using CEUS concluded that technical success was higher with Sonazoid compared to other agents .

National status: A study evaluated the role of CEUS in guiding RFA of HCC, however the contrast used was SonoVue and no comparison was made of the post op CEUS with routine 1 month imaging .

The purpose of this study is to evaluate role of perfluorobutane in guiding ablation (RFA/MWA) of HCC and to compare treatment response two hours post procedure using the same ultrasound contrast agent with routine follow up CT/MRI at 1 month post procedure.

* Why this study- Sonazoid is available in only limited countries as of now (Japan, South Korea, Norway)
* So only limited efficacy studies have been done and none in India.
* Also, no study as yet has simultaneously evaluated role of Sonazoid in both lesion targeting as well as response assessment.
* Hypothesis- Immediate post-procedure CEUS with Sonazoid is not inferior to routine contrast CT/MRI at 1 month follow-up for response assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult s (18 80 years) with HCC and who refused surgical resection
2. Tumour number not more than five and the largest tumour size not larger than 5.0 cm;
3. Ill defined lesions which are not easily detected on grey scale USG for lesion targeting.
4. Liver function status at Child Pugh class A or B;
5. East Coast Oncology Group (ECOG) performance status value 0 or 1;
6. No severe coagulopathy (e.g. platelets ≥50,000/ prothrombin time ratio ≥ 50%).
7. Available medical records and/or imaging studies.

Exclusion Criteria:

1. Presence of vascular invasion and extrahepatic metastases at pre procedure imaging study;
2. Ongoing anticoagulant treatment that cannot be stopped;
3. Combined TACE and ablation for a larger lesion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Comparison of treatment response two hours post procedure with Perfluorobutane with routine CECT/CEMRI done at 1 month post procedure using modified RECIST criteria for HCC. | upto 6 months
  Post procedure CEUS will be done which will be compared with 1 month CECT/CEMRI to compare treatment response of ablation

SECONDARY OUTCOMES:
Targeting of lesions (fulfilling CEUS LIRADS 4/5 criteria) in the Kupffer phase for ablation | upto 6 months
  Lesions will be targeted in the Kupffer phase based on their appearance in the arterial and venous appearance which should fulfil CEUS LIRADS criteria for HCC. Part of the lesion showing maximum arterial enhancement will be targeted which can include a larger area than what is seen on gray scale USG alone. This will lead to better and complete ablation of the lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Mukund, MBBS, MD, Study Director — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mukund A, Bansal A, Patidar Y, Thapar S, Sharma MK, Sarin SK. Role of contrast-enhanced ultrasound with Perfluorobutane in lesion detection, guidance for microwave ablation, and response assessment of hepatocellular carcinoma. Abdom Radiol (NY). 2022 Oct;47(10):3459-3467. doi: 10.1007/s00261-022-03609-y. Epub 2022 Jul 16. PMID 35842563